CLINICAL TRIAL: NCT00292370
Title: A Placebo-controlled Trial of Adjunctive Quetiapine for Refractory PTSD
Brief Title: Quetiapine Augmentation for Treatment-resistant PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-006-04F
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Combat Disorders; Stress Disorders, Post-Traumatic
Keywords: Atypical Antipsychotics; Controlled Trial; Paroxetine; Quetiapine; Stress Disorders, Post-Traumatic; Treatment refractory; Treatment resistant
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Paroxetine; Sugars; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Open Label (OL) Paroxetine (Other): Open-label Paroxetine In Phase I, eligible participants will take open-label (OL) Paroxetine (up to 60 mg) daily for 8 weeks. Participants who are refractory (less than 30% reduction in CAPS scores or a minimum CAPS of 50 at week 8) and have PTSD symptoms of at least moderate severity on CGI-S will be eligible for Phase II.
  Interventions: Drug: Open Label (OL) Paroxetine
- Arm 2 OL Paroxetine + DB Placebo (Placebo Comparator): In Phase II, participants will continue taking open label paroxetine and will be randomized to the addition of placebo for 8 weeks in a double-blind (DB) fashion.
  Interventions: Drug: Open Label (OL) Paroxetine; Drug: Placebo
- Arm 3: OL Paroxetine + DB Quetiapine (Experimental): In Phase II, participants will continue taking open label paroxetine and will be randomized to the addition of quetiapine (up to 800 mg daily) for 8 weeks in a double blind fashion.
  Interventions: Drug: Open Label (OL) Paroxetine; Drug: Quetiapine

INTERVENTIONS:
Drug: Open Label (OL) Paroxetine — Open-label Paroxetine
  Other Names: Paxil
Drug: Placebo — Double-blind placebo taken with OL paroxetine
  Other Names: sugar pill
  Arms: Arm 2 OL Paroxetine + DB Placebo
Drug: Quetiapine — Double-blind quetiapine taken with OL paroxetine
  Other Names: Seroquel
  Arms: Arm 3: OL Paroxetine + DB Quetiapine

SUMMARY:
The purpose of this study is to compare the response of veterans with PTSD without an optimal response to paroxetine to quetiapine augmentation versus placebo.

DETAILED DESCRIPTION:
This is a two-site study designed to evaluate the efficacy and safety of quetiapine augmentation of paroxetine treatment in veterans with PTSD who have failed to respond to paroxetine treatment.

In Phase I, eligible patients will take open-label paroxetine (up to 60 mg daily) for 8 weeks. Patients who are refractory (less than 30% reduction in CAPS scores or a minimum CAPS score of 50 at week 8) and have PTSD symptoms of at least moderate severity on CGI-S will be eligible for the second phase. In Phase II, patients will continue taking open-label paroxetine and will be randomized to the addition of quetiapine (up to 800 mg daily) or placebo for 8 weeks in a double-blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* Veteran age 18 to 75.
* Competent to give informed consent.
* Meeting DSM-IV criteria for PTSD.
* Minimal CAPS score of 50 at baseline.
* If female of childbearing potential, patient must have a negative pregnancy test and, if sexually active, be using a medically approved contraceptive method.
* Patients who have not taken psychiatric medications within 1 week prior to study entry (except fluoxetine [5 weeks])

  * monoamine oxidase inhibitors (MAOIs [4 weeks])
  * depot neuroleptics [4 weeks])
  * or any investigational drug within 30 days prior to study enrollment.
* To be eligible for Phase II

  * patients must be refractory to paroxetine in Phase I, as defined by less than 30% reduction in CAPS scores or a minimum CAPS score of 50 at week 8
  * must have PTSD symptoms at least moderate severity on CGI-S
  * and must have been compliant with study medicine in Phase I, as defined by taking at least 80% of prescribed doses.

Exclusion Criteria:

* History of sensitivity to paroxetine or quetiapine.
* Failure to respond to a prior adequate therapeutic trial i.e. minimum of 8 weeks at maximum tolerated dose of paroxetine (up to 60 mg daily) or quetiapine (up to 800 mg daily).
* Women who are

  * breast-feeding
  * pregnant
  * expect to become pregnant during the course of the study
  * or are sexually active and are not using a medically acceptable method of birth control.
* Presence of clinically significant hepatic

  * cardiovascular
  * or other medical conditions that may prevent safe administration of paroxetine or quetiapine
  * or any other clinically significant unstable medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Hamner, MD BS, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Tuscaloosa VAMC, Tuscaloosa, Alabama
  - Ralph H. Johnson, Charleston, South Carolina

REFERENCES:
- [Background] Weathers FW, Keane TM, Davidson JR. Clinician-administered PTSD scale: a review of the first ten years of research. Depress Anxiety. 2001;13(3):132-56. doi: 10.1002/da.1029. PMID 11387733
- See also: The National Center for PTSD is part of the US Department of Veterans Affairs — https://www.ptsd.va.gov/index.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1/Open-Label (OL) Paroxetine: Phase I : Open-label Paroxetine
  In Phase I, eligible participants will take open-label (OL) paroxetine (up to 60 mg daily) for 8 weeks. Participants who are refractory (less than 30% reduction in CAPS scores or a minimum CAPS score of 50 at week 8) and have PTSD symptoms of at least moderate severity on CGI-S will be eligible for Phase II
- Arm 2/OL Paroxetine & Double-blind Placebo: Phase II : Double-blind placebo
  In Phase II, participants will continue taking open-label paroxetine and will be randomized to the addition of placebo for 8 weeks in a double-blind fashion.
- Arm 3/OL Paroxetine & Double-blind Quetiapine: Phase II : Double-blind quetiapine
  In Phase II, participants will continue taking open-label paroxetine and will be randomized to the addition of quetiapine for 8 weeks in a double-blind fashion.
Period: Phase I - Open-Label Paroxetine (OLP)
Arm/Group | Arm 1/Open-Label (OL) Paroxetine | Arm 2/OL Paroxetine & Double-blind Placebo | Arm 3/OL Paroxetine & Double-blind Quetiapine
Started | 124 | 0 | 0
Completed | 78 | 0 | 0
Not Completed | 46 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Phase II: OLP + DB Quetiapine or Placebo
Arm/Group | Arm 1/Open-Label (OL) Paroxetine | Arm 2/OL Paroxetine & Double-blind Placebo | Arm 3/OL Paroxetine & Double-blind Quetiapine
Started | 0 (78 Completed Ph I 28 Excluded Ph II: * 20 responded * 7 declined * 1 medical 50 to Arm 2 & 3) | 25 (25 out of 50 in Arm I PhI, eligible for Ph II) | 25 (25 out of 50 in Arm I PhI, eligible for Ph II)
Completed | 0 | 21 | 18
Not Completed | 0 | 4 | 7
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Period 1 or Phase I, 124 patients enrolled in Arm 1/Open-Label Paroxetene for 8 weeks.
  Period 2 or Phase II (intervention period), 50 patients enrolled from week 8 to week 16; 25 in Arm 2/OL paroxetene & DB Placebo, 25 in Arm 3/OL paroxetene & DB quetiapine.
Groups:
- Arm 2/OL Paroxetine & Double-blind Placebo: Phase II: Double-blind placebo
  In Phase II, participants will continue taking open-label paroxetine and will be randomized to the addition of placebo for 8 weeks in a double-blind fashion.
- Arm 3/OL Paroxetine & Double-blind Quetiapine: Phase II: Double-blind quetiapine
  In Phase II, participants will continue taking open-label paroxetine and will be randomized to the addition of quetiapine in a double-blind fashion.
- Total: Total of all reporting groups
Arm/Group | Arm 1/Open-Label (OL) Paroxetine | Arm 2/OL Paroxetine & Double-blind Placebo | Arm 3/OL Paroxetine & Double-blind Quetiapine | Total
Number analyzed (Participants) | 124 | 25 | 25 | 174
Age, Customized [Mean (Standard Deviation); unit: years]
  Age - OL Paroxetine | 52.32 (13.23) | NA (NA) — DB participants not randomized in OL phase I (period 1) | NA (NA) — DB participants not randomized in OL phase I (period 1) | 52.32 (13.23)
  Age - Double Blind | NA (NA) — Only randomized participants counted in phase II (period 2). | 57.17 (8.74) | 54.45 (13.69) | 54.76 (11.48)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Gender for Open - Label (OL) population. Double-Blind participants not randomized in OL Phase.
  Participants
    Gender OL Females: number analyzed (Participants) | 124 | 0 | 0 | 124
    Gender OL Females | 5 |  |  | 5
    Gender OL Males: number analyzed (Participants) | 124 | 0 | 0 | 124
    Gender OL Males | 119 |  |  | 119
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Gender for Double-Blind phase II
  Participants
    Females Double Blind: number analyzed (Participants) | 0 | 25 | 25 | 50
    Females Double Blind | 0 | 1 | 1 | 2
    Males Double Blind: number analyzed (Participants) | 0 | 25 | 25 | 50
    Males Double Blind | 0 | 24 | 24 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity for Open-Label Phase participants
  Participants
    OL Amer Indian/ Alask Native: number analyzed (Participants) | 124 | 0 | 0 | 124
    OL Amer Indian/ Alask Native | 2 |  |  | 2
    OL African American: number analyzed (Participants) | 124 | 0 | 0 | 124
    OL African American | 50 |  |  | 50
    OL White: number analyzed (Participants) | 124 | 0 | 0 | 124
    OL White | 68 |  |  | 68
    OL Unknown or Not Reported: number analyzed (Participants) | 124 | 0 | 0 | 124
    OL Unknown or Not Reported | 4 |  |  | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity for Double-Blind participants
  Participants
    DB Amer Indian/ Alaska Native: number analyzed (Participants) | 0 | 25 | 25 | 50
    DB Amer Indian/ Alaska Native |  | 0 | 0 | 0
    DB African American: number analyzed (Participants) | 0 | 25 | 25 | 50
    DB African American |  | 15 | 10 | 25
    DB White: number analyzed (Participants) | 0 | 25 | 25 | 50
    DB White |  | 9 | 14 | 23
    DB Unknown/ Not Reported: number analyzed (Participants) | 0 | 25 | 25 | 50
    DB Unknown/ Not Reported |  | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants] — Population: Same region as in OL phase
  Participants
    United States: number analyzed (Participants) | 124 | 0 | 0 | 124
    United States | 124 |  |  | 124
Years of Education [Mean (Standard Deviation); unit: years]
  Education - Open Label (OL) Population | 13.12 (2.05) | NA (NA) — DB participants not yet randomized in OL, phase I. | NA (NA) — DB participants not yet randomized in OL, phase I. | 13.12 (2.05)
  Education - Double Blind (DB), Phase II | NA (NA) — Only randomized participants counted in DB, phase II. | 13.22 (2.74) | 12.55 (1.53) | 12.89 (2.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale for DSM-IV Total Score.
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS) is described in the National Center for PTSD Instruction Manual (November 2000) as a semi-structured clinical interview designed to assess the seventeen symptoms for Post Traumatic Stress Disorder (PTSD) outlined in the DSM-IV, along with five associated features. Ratings are made on a 5 point continuum from the lowest frequency or intensity to the highest. Total CAPS score is a summed score that ranges from 0 to 136 where 0 is asymptomatic and higher scores equal more severe PTSD symptomatology. Also, a change in total CAPS score of 15 points was proposed as clinically significant change.
Time Frame: From baseline (week 8) to endpoint (week 16 or termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  CAPS Total Baseline | 72.15 (15.96) | 68.78 (17.01)
  CAPS Total Endpoint | 67.90 (14.90) | 51.52 (19.68)
Statistical Analysis 1: Comparison: Arm 2 OL Paroxetine + DB Placebo vs Arm 3: OL Paroxetine + DB Quetiapine; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in CGI-I
Description: Clinical Global Impressions Scale and Global Improvement Subscales (CGI-I) is a 7-point scale which was used to assess overall improvement. The scores range from 1 to 7, with 1 indicating very much improved and 7 indicating very much worse.
Time Frame: From Baseline (week 8) to Endpoint (week 16 or termination)
Population: Randomized participants with CGI-I score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline CGI-I | 3.56 (.85) | 3.36 (.88)
  Endpoint CGI-I | 2.61 (.79) | 2.22 (1.19)

3. Secondary Outcome: Change in Mean PANSS Total and Subscores From Baseline to Endpoint
Description: Positive and Negative Symptom Scale (PANSS). A 30-item clinician administered rating scale for which positive, negative and general subscales are scored from 30 to 210 with a higher scores indicating greater severity of symptoms.
Time Frame: Baseline (week 8) to Endpoint (week 16 or termination)
Population: Randomized participants with a PANSS score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline Total PANSS | 46.63 (10.13) | 47.76 (11.09)
  Endpoint Total PANSS | 43.92 (6.81) | 42.24 (8.07)

4. Secondary Outcome: Change in Total Mean Hamilton Rating Scale for Depression (HAMD) Scores
Description: Hamilton Rating Scale for Depression (HAMD) was used as a measure of depression. Scoring is based on a 17-item scale. Eight items are scored on a 5 point scale from 0= not present to 4= severe. The scoring is based on the first 17 items. Scores of 0-7 normal, 8-13 is mild depression, 14-18 moderate depression, 19-22 severe depression and 23 and above very severe depression; the maximum score being 52 on the 17-point scale.
Time Frame: From Baseline (week 8) to Endpoint (week 16 or Termination)
Population: Randomized participants with a HAMD score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline HAMD | 14.60 (5.45) | 13.84 (6.05)
  Endpoint HAMD | 12.29 (6.35) | 9.29 (4.56)

5. Secondary Outcome: Change in Total Mean Davidson Trauma Scale (DTS)
Description: The DTS is a 17-item self-rated scale that measures the frequency and the severity of DSM-IV PTSD symptoms. Items are rated on 5-point frequency (0 = "not at all" to 4 = "every day") and severity scales (0 = "not at all distressing" to 4 = "extremely distressing"). The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). A higher score indicates higher frequency and severity. It can be used to make a preliminary determination about whether the symptoms meet DSM criteria for PTSD. Scores can also be calculated for each of the 3 PTSD symptom clusters (i.e., B, C, and D).
Time Frame: From Baseline (week 8) to Endpoint (week 16 or Termination)
Population: Randomized participants with a DTS score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline DTS | 82.19 (24.60) | 77.25 (25.94)
  Endpoint DTS | 84.06 (21.92) | 61.50 (18.20)

6. Secondary Outcome: Change in Mean Q-LES-Q Score From Baseline to Endpoint.
Description: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) a self-rated 14-item questionnaire designed to assess the degree of enjoyment and satisfaction of various aspects of daily functioning. Each question is rated on a 5-point scale with scores ranging from "1 = very poor" to "5 = very good". The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70. A lower score indicates worsening and a higher score indicates better quality of life.
Time Frame: From Baseline (week 8) to Endpoint (week 16 or termination)
Population: Randomized participants with a Q-LES-Q score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline Q-LES-Q | 37.85 (7.78) | 40.44 (8.82)
  Endpoint Q-LES-Q | 38.22 (6.62) | 41.06 (6.70)

7. Secondary Outcome: Change in Mean Scores of Pittsburgh Sleep Quality Index (PSQI) From Baseline to Endpoint.
Description: The PSQI is one of the most frequently used self-rated sleep questionnaire. Total score ranging from 0 to 21. Higher scores are representing worse sleep quality.
Time Frame: From Baseline (week 8) to Endpoint (week 16)
Population: Randomized participants with a PSQI score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline PSQI | 11.60 (3.93) | 12.69 (3.46)
  Endpoint PSQI | 8.70 (3.15) | 13.19 (2.88)

8. Secondary Outcome: Change in Mean Sheehan Disability Scale (SDS) Scores From Baseline to Endpoint.
Description: The SDS is a brief 3-item questionnaire that was used as a self-report to assess the degree to which psychiatric symptoms have disrupted the patient's work, family/home responsibilities, and social life. Score ranging from 0 (no impairment) to 30 (most severe).
Time Frame: Baseline (week 8) to Endpoint (week 16 or termination)
Population: Randomized participants with an SDS score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline SDS-WS | 5.07 (3.45) | 4.44 (2.95)
  Endpoint SDS-WS | 4.58 (2.99) | 4.66 (2.34)
  Baseline SDS-SL | 6.67 (2.44) | 5.64 (2.93)
  Endpoint SDS-SL | 5.92 (2.55) | 4.95 (1.83)
  Baseline SDS-FL | 5.85 (2.92) | 4.72 (2.48)
  Endpoint SDS-FL | 5.39 (2.48) | 4.61 (2.27)

9. Secondary Outcome: Change in Arizona Sexual Experience Scale (ASEX)
Description: The ASEX is a brief 5-item rating scale that assesses five global aspects of sexual dysfunction. Score is 5 and the maximum score is 30. Lower scores indicate more positive sexual experiences.
Time Frame: From Baseline (week 8) to Endpoint (week 16 or termination)
Population: Randomized participants with an ASEX score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline ASEX | 22.00 (6.68) | 17.88 (5.33)
  Endpoint ASEX | 21.93 (7.45) | 16.94 (5.84)

ADVERSE EVENTS:
Time Frame: Collected over 4 months per subject.
Description: Collected by open-ended questions, vitals, standardized report form, and chart review at visits every two weeks, as well as by lab assessments between phases I and II.
Groups:
- Arm 1: Open Label (OL) Paroxetine: In Phase I, eligible participants will take open-label (OL) Paroxetine (up to 60 mg) daily for 8 weeks. Participants who are refractory (less than 30% reduction in CAPS scores or a minimum CAPS of 50 at week 8) and have PTSD symptoms of at least moderate severity on CGI-S will be eligible for Phase II.
  Open Label (OL) Paroxetine: Open-label Paroxetine
Arm/Group | Arm 1: Open Label (OL) Paroxetine | Arm 2 OL Paroxetine + DB Placebo | Arm 3: OL Paroxetine + DB Quetiapine
Serious Adverse Events (participants affected / at risk) | 5/124 | 0/25 | 2/25
Other Adverse Events (participants affected / at risk) | 23/124 | 2/25 | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Open Label (OL) Paroxetine (N=124) | Arm 2 OL Paroxetine + DB Placebo (N=25) | Arm 3: OL Paroxetine + DB Quetiapine (N=25)
Hospitalized - Suicide Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — suicide Ideation and substance abuse
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) — Hypotension
Hospitalized - scheduled cardiac stint (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) — Scheduled cardiac stint
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Open Label (OL) Paroxetine (N=124) | Arm 2 OL Paroxetine + DB Placebo (N=25) | Arm 3: OL Paroxetine + DB Quetiapine (N=25)
Sexual Side effects (Reproductive system and breast disorders) | 10 (10) | 1 (1) | 1 (1) — sexual dysfunction
Sedation (Nervous system disorders) | 7 (7) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Heart palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No